CLINICAL TRIAL: NCT07206693
Title: Impact of PSA-based Screening on Mortality Among Men Aged 75-79: Target Trial Emulation
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Tobias Nordström, MD PhD, Karolinska Institutet
Other Study IDs: 2012/438-31/3
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Prostate Cancer Screening; Prostate Cancer Screening Decision; Prostate Specific Antigen Screening
Keywords: prostate cancer; screening; prostate specific antigen; older adults; urology; mortality; emulation of target trial
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 17 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men aged 75-79 living in Stockholm from 2007-2023
  Interventions: Diagnostic Test: Prostate specific antigen (PSA)

INTERVENTIONS:
Diagnostic Test: Prostate specific antigen (PSA) — Prostate specific antigen (PSA) for prostate cancer screening

SUMMARY:
Opportunistic prostate-specific antigen (PSA) testing is widespread among men aged 75-79. Current American and European guidelines recommend PSA-based screening through shared decision-making if men are expected to live at least 10 more years-a threshold previously tied to ages 70-74. With rising life expectancy, Swedish men aged 75-79 now exceed this benchmark, averaging over 10 years.

Since no randomized controlled trials have examined screening in this age group, this study will use data from the Stockholm Prostate Cancer Diagnostics Register (2007-2023) to emulate a target trial. Men without prior prostate cancer will be assigned to screened or unscreened groups based on PSA test records and followed until death or December 2023. Analyses will use survival models, cumulative incidence functions, and sensitivity checks (e.g., varying follow-up duration, calendar year vs. age enrollment, and comparisons with men aged 65-69).

The goal is to determine whether PSA screening at ages 75-79 improves overall and prostate cancer-specific survival, and whether guidelines should expand to include this group while balancing the risk of overdiagnosis. Results will inform both clinical practice and the design of future randomized trials.

ELIGIBILITY:
Inclusion Criteria:

Men aged 75-79 between 2007-2023, with no prostate cancer diagnosis at the time of inclusion (based on each trial emulation) will be considered eligible for the trials. To ensure proper control for potential confounding, and to be able to evaluate the eligibility criteria, only men with complete information on their screening status, outcomes, and confounders in the registers will be included.

Exclusion Criteria:

Men younger than 75 or older than 79 between 2007-2023. Have prostate cancer diagnosis at the time of inclusion (based on each trial emulation) Missing data on the exposure, outcomes, and confounders.

Ages: 75 Years to 79 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study and the target-trial emulation will use population-based register data of men living in Stockholm between 2007-2023 screened for prostate cancer, extracted from the Stockholm Prostate Cancer Diagnostics Register (STHLM0). STHLM0 has complete PSA test records since 1 January 2007. This will be supplemented with information on non-tested men from the STHLM0+ register. Demographic information, family history of prostate cancer, diagnoses, hospitalization, specialized outpatient healthcare, prostate cancer treatment, and mortality information are provided from the linked Swedish population registers
Sampling Method: Non-Probability Sample
Enrollment: 257275 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 17 years
Prostate-cancer specific mortality | 17 years

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Nordström, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared publically because of restrictions from Swedish laws and GDPR. However, the IPD can be requested from the study PI following approval from the Swedish ethics committee, and approval of the data sharing agreement between the two institutions at Karolinska Institutet.

REFERENCES:
- [Derived] Abbadi A, Micoli C, Discacciati A, Olarte Parra C, Lantz A, Bjornebo L, Arvendell M, Chandra Engel J, Andersson J, Falagario U, Gronberg H, Eklund M, Clements M, Nordstrom T. Can Prostate Cancer Screening Reduce Mortality in Men Aged 75-79 Years? A Protocol for Target-trial Emulation. Eur Urol Open Sci. 2025 Nov 6;82:147-154. doi: 10.1016/j.euros.2025.10.016. eCollection 2025 Dec. PMID 41280154